CLINICAL TRIAL: NCT04144621
Title: The Correlation of Sperm DNA Fragmentation With Blastocyst Grading and Its Implantation Potential
Brief Title: Sperm DNA Fragmentation Effects on Blastocyst Morphology Grading, Pregnancy Rate and Implantation Rate
Status: Completed | Type: Observational
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Sponsor
Other Study IDs: MH0001
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Blastocyst; Implantation Rate
Keywords: Sperm DNA fragmentation; Implantation rate; Pregnancy rate; Blastocyst grading
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — semen, oocytes, blastocysts
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal SDF: Couples with male partners having SDF lower than 20% using TUNEL assay
  Interventions: Procedure: ICSI
- Abnormal SDF: Couples with male partners having SDF greater than 20% using TUNEL assay
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — Intracytoplasmic sperm injection of female partner oocytes with ejaculated sperm selected by density gradient centrifugation

SUMMARY:
Retrospective cohort study for 189 couples assigned to normal and abnormal Sperm DNA fragmentation (SDF) groups.To determine the effect of SDF on blastocyst's trophectoderm (TE), Inner cell mass (ICM) morphology grading, and implantation rate. Semen in both groups was processed by density gradient (DG).

DETAILED DESCRIPTION:
Purpose: to determine if sperm DNA fragmentation (SDF) has a correlation with Blastocyst's trophectoderm (TE) and Inner cell mass (ICM) grading, or with the implantation rate?

Method: Retrospective cohort study for 189 couples, assigned to normal SDF group (121 cases), and abnormal SDF group (68 cases). Semen in both groups was processed by double layer density gradient (DG).

Statistical analysis done using SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* All cases in this study have to reach the blastocyst stage.
* Female age ≤37 years old.
* Male sperm count ≥ 5 million.

Exclusion Criteria:

* Usage of sperm selection techniques.
* Testicular aspiration or testicular biopsies.
* Oocyte or sperm donation.

Max Age: 37 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes — female age ≤37 years old, with no limitation on male age
Study Population: ICSI patients in Ganin Fertility Center from January 2018 to September 2018.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Blastocyst morphological grading | 5-6 days after ICSI
  Morphological grading of trophectoderm and Inner cell mass using Gardner's criteria 1999, from grade A to C ( A is the highest quality).
Implantation rate | 6 weeks of pregnancy
  Percentage of the implanted embryos number for each group / number of transferred embryos.

SECONDARY OUTCOMES:
Fertilization rate | 16-19 hours of ICSI
  Percentage of fertilized oocyte (appearance of two pronuclei) / Number of injected oocytes
Blastulation rate | 5-6 days of ICSI
  Percentage of total blastocysts / total 2PN
Pregnancy rate | After 2 weeks of embryo transfer
  Percentage of pregnant cases / transferred cases for each group ( positive pregnancy test)

CONTACTS AND LOCATIONS:
Overall Officials: Manar Hozyen, MSc, Principal Investigator — Ganin Fertility Center; Eman Hassanen, BSc, Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc, FRCOG, Study Chair — Ganin Fertility Center; Hanaa El Khedr, Principal Investigator — Ganin Fertility Center; Yasmine Azzouz, BSc, Principal Investigator — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Egypt

REFERENCES:
- [Background] Wdowiak A, Bojar I. Relationship between pregnancy, embryo development, and sperm deoxyribonucleic acid fragmentation dynamics. Saudi J Biol Sci. 2016 Sep;23(5):598-606. doi: 10.1016/j.sjbs.2015.08.001. Epub 2015 Aug 10. PMID 27579009
- [Background] Gat I, Tang K, Quach K, Kuznyetsov V, Antes R, Filice M, Zohni K, Librach C. Sperm DNA fragmentation index does not correlate with blastocyst aneuploidy or morphological grading. PLoS One. 2017 Jun 7;12(6):e0179002. doi: 10.1371/journal.pone.0179002. eCollection 2017. PMID 28591199
- [Background] Alvarez Sedo C, Bilinski M, Lorenzi D, Uriondo H, Noblia F, Longobucco V, Lagar EV, Nodar F. Effect of sperm DNA fragmentation on embryo development: clinical and biological aspects. JBRA Assist Reprod. 2017 Dec 1;21(4):343-350. doi: 10.5935/1518-0557.20170061. PMID 29116706